CLINICAL TRIAL: NCT01997476
Title: Evaluation of Combined Endoscopic Ultrasound Ductal Evaluation Before & After Secretin Stimulation in One EUS Session for the Diagnosis of Exocrine Pancreas Disease
Brief Title: EUS Ductal Evaluation in One Endoscopic Session for the Diagnosis of Exocrine Pancreas Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Director of Endosocpic Ultrasound, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1105005314/1010-26
Record Dates: First submitted 2013-11-13; First posted 2013-11-28 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Pancreatic Disease
Keywords: Combined Endoscopic Ultrasound Morphologic Evaluation.
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined EUS, e-PFT and sEUS Testing (Experimental): Establish the advantage of combined EUS, ePFT & sEUS testing to provide a more definitive diagnostic assessment, rather than each test alone.
  Establish the advantage of reduced time and cost of combining EUS and ePFT, rather than when done separately.
  Interventions: Procedure: Combined EUS, e-PFT and sEUS Testing

INTERVENTIONS:
Procedure: Combined EUS, e-PFT and sEUS Testing — advantage of combined EUS, ePFT & sEUS testing to provide a more definitive diagnostic assessment, rather than each test alone.
  Establish the advantage of reduced time and cost of combining EUS and ePFT, rather than when done separately.

SUMMARY:
The purpose of this study is, to develop a standard of care protocol using the combination of EUS, ePFT, and sEUS during one endoscopic session (instead of the three separate endoscopic sessions). The desired outcome is to diagnose CP and to establish an acceptable protocol for performing this combined technique. It is expected that combining these procedures will eliminate redundant portions of the procedures, reduce repeat visits to the hospital, reduce total recovery time for the patient, and will decrease the associated costs of separate procedures. Chronic pancreatitis (CP) is an irreversible, disease in which the pancreas becomes fibrotic ( thickened and scarred). Symptoms almost always include pain, and as the pancreas becomes progressively more fibrosed (thickened), pancreatic hormonal function is compromised with diarrhea and weight loss. However, while most physicians can readily diagnose patients with severe CP, early CP or "minimal-change" CP is difficult to detect, often due to the lack of radiologic findings, laboratory tests and classic symptoms. As a result, clinicians are searching for diagnostic tools which will allow for earlier, accurate detection of this disease, with the hope that appropriate therapy can be initiated before extensive thickening and scarring of the pancreas occurs.

Diagnostic tools to evaluate the pancreas include Endoscopic Ultrasound (EUS), hormone-stimulated endoscopic pancreatic function tests (ePFT) and Secretin stimulated Endoscopic Pancreas Function Test (sPFT) using pancreatic fluid (containing bicarbonate) obtained from the duodenum (the part of the intestine where the stomach opens into the small bowel). EUS is increasingly being used as a diagnostic and treatment tool in pancreatic disease. Currently, hormone-stimulated ePFT is considered the best way to diagnose chronic pancreatitis (long-lasting inflammation and scarring of the pancreas), and removes the need for biopsy or surgery. It is also sensitive in detecting mild disease.

These procedures are standard of care (the normal care you would receive) for the evaluation of CP. The purpose of this study, is to develop a standard of care protocol using the combination of EUS, ePFT, and sEUS during one endoscopic session, instead of three separate endoscopic procedures.

DETAILED DESCRIPTION:
Combined EUS, e-PFT and sEUS Testing:

The endoscopic procedures for this study will be performed by a single endoscopist at each center. It is expected that the combined EUS, ePFT and sEUS will be completed in less than 75 minutes. Patient sedation will be accomplished via standard conscious (Midazolam, Fentanyl and/or Meperidine) sedation or monitored (Propofol) sedation as per the study investigator and America Society of Gastrointestinal Endoscopy (ASGE) and American Society of Anesthesiology (ASA) guidelines.

A mechanical-radial EUS echoendoscope with color Doppler assessment capability will be passed via standard technique and the pancreas examined from the gastric and duodenal stations. Representative EUS images will be recorded on digital videotape/digital snapshot from the head, body and tail per the CRF. See Appendix B. These images will then become part of the patient's electronic medical record. The echoendoscope will be used to measure specific parenchymal (hyperechoic foci with shadowing, hyperechoic strands with shadowing, lobular contour, cysts, calculi) and ductal (main ductal diameter, irregularity, hyperechoic margins, stones and the presence of visible side branches) abnormalities. It is expected that this evaluation will be completed in approximately 10 minutes. Prior to secretin administration (baseline MPD diameters), the pancreatic duct diameter will be measured in the head, body, and tail using endosonographic calipers. The investigator will provide an initial assessment of the presence or absence of chronic pancreatitis prior to secretin administration.

Next, the echoendoscope will be used to aspirate the gastric and duodenal lumens dry. The gastric and duodenal samples will then be discarded.

Once the gastric and duodenal lumens have been aspirated dry, patients will be given a test dose of human secretin of 0.2 mcg (0.1mL) through an indwelling catheter in a peripheral vein to assess for a possible allergic response. Patients will be monitored at all times for evaluation of hemodynamic instability. If after one minute there is no evidence of an allergic reaction, the remaining full dose of secretin 0.2 mcg/kg IV will be given over one minute.

Beginning at time 4 minutes after the completion of secretin intravenous infusion, the pancreatic duct diameter will be measured in the head, body, and tail using endosonographic calipers. Measurements of the pancreatic duct will occur sequentially at 4, 8, and 12 minutes following the conclusion of secretin administration. Representative images will also be obtained of each measurement at each time point. The echoendoscope will be used to measure specific parenchymal (hyperechoic foci with shadowing, hyperechoic strands with shadowing, lobular contour, cysts, calculi) and ductal abnormalities. The investigator will perform a follow-up assessment of chronic pancreatitis using additional data on post-secretin administration.

The ePFT portion of the examination will then commence. The echoendoscope will be removed and a forward-viewing gastroscope placed into the stomach. Stomach contents will then be aspirated dry. The forward-viewing gastroscope will then be placed across the pylorus into the distal duodenum. Beginning time 15 minutes following the completion of the secretin infusion, duodenal samples (5-10 mL) will be collected through the suction channel of the echoendoscope. The samples will be collected in a standard endoscopic collection container and placed on ice. At time 30 and 45 minutes after the completion of secretin administation, samples will obtained in a similar fashion and placed in separate containers on ice. The procedure will then be completed and the patient brought to the same day recovery suite.

At the conclusion of the procedure, the samples will be brought immediately to the hospital chemistry laboratory where they will be evaluated for bicarbonate concentration using the hospital autoanalyzer or frozen at -70 degrees Celsius if analysis is delayed. Using the autoanalyzer for this technique generally requires a three-fold dilution of the fluid contents. The highest bicarbonate concentration from the 3 samples will be considered the peak concentration. The diagnostic cut-off for pancreatic exocrine disease will be set at < 80 mEq/L (80 mEq/L or greater indicates normal function).

Patient participation in the study will be completed at the time of completion of their combined function testing. A telephone call will occur by the PI or designee to each patient within 3-7 days of study drug administration will serve as follow-up and complete the CRF.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between the ages of 18-80 years old.
2. Clinical suspicion of pancreatic exocrine disease.
3. If female and not more than 1 year post-menopausal or surgically sterile, must use medically acceptable form of contraception or abstain from sexual activity during the study. Acceptable methods of birth control are: intrauterine device, implantable progesterone device, progesterone intramuscular injection, oral contraceptive (started at least one month prior to Screening Visit 1 and continuing for the duration of the trial), contraceptive patch, condoms with spermicide or abstinence.
4. EUS and ePFT planned for structural and functional evaluation of the exocrine pancreas.
5. Ability to undergo conscious sedation or monitored anesthesia.
6. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Symptoms of acute pancreatitis within 30 days of the combined function test.
2. Severe cardiac disease (stable or unstable angina, congestive heart failure, uncontrolled arrhythmias, implantable defibrillator, severe valvular disease, etc).
3. Severe pulmonary disease (COPD, severe asthma, interstitial lung disease, etc).
4. Severe renal disease (history of acute or chronic renal failure and/or dialysis dependent and/or baseline creatinine >2.0 mg/dL).
5. Pregnant or nursing.
6. Ongoing illicit drug use or abuse.
7. Ongoing moderate or severe alcohol use defined by greater than 30 grams alcohol/day.
8. Acute pancreatitis as defined by the Atlanta Classification definition (see Appendix D) within the previous two months.
9. Prior pancreatic surgery.
10. Presence of a condition which may interfere with exocrine pancreatic functioning including celiac disease, type I diabetes mellitus, previous gastrectomy, cystic fibrosis or severe malnutrition (BMI <18).
11. Exhibiting signs or symptoms of an episode of acute pancreatitis.
12. Known allergy to secretin.
13. Recent (within 30 days) use of medication that can potentially cause pancreatitis, such as metronidazole, tetracycline, sulfonamides.
14. Use of any anticholinergic medication within 48 hours of enrollment.
15. Any medical condition which in the judgment of the Investigator renders participation in this study medically inadvisable.
16. Participation in an investigational clinical study for a drug or medical device within 30 days prior to Screening Visit 1.
17. Suspected or proven Sphincter of Oddi Dysfunction.
18. Previous pancreatic endoscopic or surgical sphincterotomy

    -

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Combined Endoscopic Ultrasound Morphologic Evaluation, Endoscopic Pancreatic Function Testing (ePFT), and Dynamic EUS Ductal Evaluation (sEUS) | 48 months (anticipated)
  Combined Endoscopic Ultrasound Morphologic Evaluation, Endoscopic Pancreatic Function Testing, and Dynamic EUS Ductal Evaluation before and after Human Secretin Stimulation in one Endoscopic Session for the Diagnosis of Exocrine Pancreas Disease

SECONDARY OUTCOMES:
Advantage of combining EUS and ePFT to provide a more definitive diagnostic assessment, rather than each test alone. | 48 months (anticipated).
  Establish the advantage of combining EUS and ePFT to provide a more definitive diagnostic assessment, rather than each test alone.
  Establish the advantage of reduced time and cost of combining EUS and ePFT, rather than when done separately.

CONTACTS AND LOCATIONS:
Overall Officials: John M. DeWitt, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University; University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeWitt JM, Al-Haddad MA, Easler JJ, Sherman S, Slaven J, Gardner TB. EUS pancreatic function testing and dynamic pancreatic duct evaluation for the diagnosis of exocrine pancreatic insufficiency and chronic pancreatitis. Gastrointest Endosc. 2021 Feb;93(2):444-453. doi: 10.1016/j.gie.2020.06.029. Epub 2020 Jun 17. PMID 32562609